CLINICAL TRIAL: NCT03279796
Title: Autologous Adipose-derived Mesenchymal Stem Cells in the Treatment of Tendon Disease: a Randomized Controlled Trial
Brief Title: Treatment of Tendon Disease Using Autologous Adipose-derived Mesenchymal Stem Cells
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Zhejiang Xingyue Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017.No.55
Record Dates: First submitted 2017-09-04; First posted 2017-09-12 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2017-08

CONDITIONS: Rotator Cuff Tear; Lateral Epicondylitis
Keywords: Adipose-drived mesenchymal stem cells; Rotator cuff injury; Lateral Epicondylitis; Randomized controlled trials
MeSH Terms: conditions — Rotator Cuff Injuries; Tennis Elbow

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autologous adipose-derived MSCs (Experimental): The dose of adipose-derived mesenchymal stem cells was related to body weight, and 1 × 10 ^ 6 cells were a unit. One unit of adipose-derived mesenchymal stem cells was injected every 10 kg of body weight and injected once a week for three times.
  Interventions: Biological: Autologous adipose-derived MSCs
- Compound betamethasone (Active Comparator): 1ml dexamethasone mixed with 0.5-2ml of saline to achieve the same injection volume with the cell suspension (which contains betamethasone dipropionate 5mg and betamethasone sodium phosphate 2mg) ), once a week for three times.
  Interventions: Drug: Compound betamethasone

INTERVENTIONS:
Biological: Autologous adipose-derived MSCs — The dose of adipose-derived mesenchymal stem cells was related to body weight, and 1 × 10 ^ 6 cells were a unit. One unit of adipose-derived mesenchymal stem cells was injected every 10 kg of body weight and injected once a week for three times.
  Arms: Autologous adipose-derived MSCs
Drug: Compound betamethasone — 1ml dexamethasone mixed with 0.5-2ml of saline to achieve the same injection volume with the cell suspension (which contains betamethasone dipropionate 5mg and betamethasone sodium phosphate 2mg) ), once a week for three times.
  Arms: Compound betamethasone

SUMMARY:
This study was a single-center, randomized, single-blind clinical trial. We plan to include 100 patients who met exclusion criteria of rotator cuff and lateral epicondylosis (tennis elbow) respectively by MRT or ultrasonography. The patients will be randomly divided into two groups. Adipose mesenchymal stem cells will be isolated from adipose tissue, cultured and then transplanted back to the tendon injury site by multiple point injection. 1*10^6 cells as an unit. Patients in the experiment group will be injected into an unit of adipose mesenchymal stem cells (1*10^6/10kg) while the control group received the same dose compound betamethasone injection. Follow up visit for all patients will occur at 1，3，6 and 12 months after the first injection. Clinical quantitative assessment will measure by the visual analogue scale(VAS). The secondary outcomes are the constant-murley score(CMS) and the rating scale of the American shoulder and elbow surgeons(ASES) and the disability of arm shoulder and hand(DASH). The objective evaluation methods is that the examination of MRI or ultrasound were accomplished before the first injection and at 6 and 12 months afterwards.

DETAILED DESCRIPTION:
All injection will be done under ultrasound guidance.

ELIGIBILITY:
Inclusion Criteria:

1. clinically diagnosed as rotator cuff tear or lateral epicondylitis (tennis elbow);
2. symptom duration is over 3 months, non-steroidal drug treatment , rehabilitation treatment and other conservative treatment is invalid;
3. patient that can understand the clinical trials and signed the informed consent.

Exclusion Criteria:

1. patient that underwent other injection treatment within 6 weeks
2. some associated diseases (such as arthritis, synovitis, entrapment of related nerve, radiculopathy to the target lesion, generalized pain syndrome, rheumatoid arthritis, pregnancy, impaired sensibility, paralysis, history of allergic or hypersensitive reaction to bovine-derived proteins or fibrin glue)
3. patient that enrolled other clinical trials within 3 months
4. history of drug/alcohol addiction, habitual smoker

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Visual Analog Scale(VAS) at 3, 6 and 12 weeks | Baseline, 3 weeks, 6 weeks, 12 weeks after intervention
  Pain on activity will be evaluated by VAS

SECONDARY OUTCOMES:
Change from baseline in Constant-Murley Score(CMS) at 3, 6 and 12 weeks, | Baseline, 3 weeks, 6 weeks, 12 weeks after intervention
  Functional score of the shoulder
American Shoulder and Elbow Surgeons (ASES) Shoulder Score | Baseline, 3 weeks, 6 weeks, 12 weeks after intervention
  Functional score of the shoulder
The Disabilities of the Arm, Shoulder and Hand(DASH) Score | Baseline, 3 weeks, 6 weeks, 12 weeks after intervention
  Functional score of the shoulder
Adverse events | From baseline through study completion, an average of 1 year
  Adverse events to evaluate the safety

CONTACTS AND LOCATIONS:
Locations (1):
- Weiliang Shen, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ellera Gomes JL, da Silva RC, Silla LM, Abreu MR, Pellanda R. Conventional rotator cuff repair complemented by the aid of mononuclear autologous stem cells. Knee Surg Sports Traumatol Arthrosc. 2012 Feb;20(2):373-7. doi: 10.1007/s00167-011-1607-9. Epub 2011 Jul 20. PMID 21773831
- [Background] Pascual-Garrido C, Rolon A, Makino A. Treatment of chronic patellar tendinopathy with autologous bone marrow stem cells: a 5-year-followup. Stem Cells Int. 2012;2012:953510. doi: 10.1155/2012/953510. Epub 2011 Dec 18. PMID 22220180
- [Background] Hernigou P, Flouzat Lachaniette CH, Delambre J, Zilber S, Duffiet P, Chevallier N, Rouard H. Biologic augmentation of rotator cuff repair with mesenchymal stem cells during arthroscopy improves healing and prevents further tears: a case-controlled study. Int Orthop. 2014 Sep;38(9):1811-8. doi: 10.1007/s00264-014-2391-1. Epub 2014 Jun 7. PMID 24913770
- [Background] Pas HIMFL, Moen MH, Haisma HJ, Winters M. No evidence for the use of stem cell therapy for tendon disorders: a systematic review. Br J Sports Med. 2017 Jul;51(13):996-1002. doi: 10.1136/bjsports-2016-096794. Epub 2017 Jan 11. PMID 28077355
- [Background] Lee SY, Kim W, Lim C, Chung SG. Treatment of Lateral Epicondylosis by Using Allogeneic Adipose-Derived Mesenchymal Stem Cells: A Pilot Study. Stem Cells. 2015 Oct;33(10):2995-3005. doi: 10.1002/stem.2110. Epub 2015 Aug 6. PMID 26202898
- [Background] Ouyang HW, Goh JC, Thambyah A, Teoh SH, Lee EH. Knitted poly-lactide-co-glycolide scaffold loaded with bone marrow stromal cells in repair and regeneration of rabbit Achilles tendon. Tissue Eng. 2003 Jun;9(3):431-9. doi: 10.1089/107632703322066615. PMID 12857411
- [Background] Minagawa H, Yamamoto N, Abe H, Fukuda M, Seki N, Kikuchi K, Kijima H, Itoi E. Prevalence of symptomatic and asymptomatic rotator cuff tears in the general population: From mass-screening in one village. J Orthop. 2013 Feb 26;10(1):8-12. doi: 10.1016/j.jor.2013.01.008. eCollection 2013. PMID 24403741